CLINICAL TRIAL: NCT05946187
Title: Getting Back on Track: Alternative Healthcare Delivery Strategies to Prevent Weight Regain After Bariatric Surgery
Brief Title: Alternative Healthcare Delivery Strategies to Prevent Weight Regain After Bariatric Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Collaborators: Hospital de Braga (Other); Fundação para a Ciência e a Tecnologia (Other); Centro Hospitalar De São João, E.P.E. (Other); Universidade do Porto (Other)
Responsible Party: Principal Investigator, Eva Conceição, Professor, Principal Investigator, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UMinho_ApoloBari_FB
Record Dates: First submitted 2023-05-24; First posted 2023-07-14 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Obesity Adult Onset; Eating Behavior
Keywords: alternative healthcare strategies; weight regain; eating behaviors; bariatric surgery
MeSH Terms: conditions — Feeding Behavior | interventions — Therapeutics; Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial will compare two groups: a Treatment As Usual control group with an Stepped-care intervention group. The Stepped-care approach organizes interventions with two different intensities (Steps 1-2), delivered entirely via private groups on Facebook®. A logarithm will guide when patients move to another step based on the presence of certain key symptoms. Participants will be recruited at the São João Hospital Center and at the Hospital of Braga. All participants will be contacted by the researcher after their medical appointment. Patients meeting the criteria will be invited to participate in the study and sign an informed consent form. Objectives and procedures of the investigation will be explained. The study will be introduced as a program to support bariatric patients in the long term in different modalities, which aims to monitor relevant variables and investigate patients' perceptions of the utility of these interventions.
Who Masked: Outcomes Assessor
Masking Description: Randomization is performed by a researcher not involved in data management. The researcher who evaluates the outcomes of interest is masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apolo_Bari Stepped-care intervention group (Experimental): The Apolo_Bari stepped-care intervention offers two different steps from low- to high-intensity strategies. The intervention will run for 18 months. All participants receive first step intervention. Patients will move through the second step according to the degree of disordered eating behaviors or weight regain which is assessed through a short Monthly Monitoring Questionnaire.
  Interventions: Behavioral: Apolo_Bari Stepped-care intervention
- Treatment as usual group (Active Comparator): Treatment As Usual control group receives the standard intervention for bariatric surgery offered by multidisciplinary teams in Portuguese public hospitals. It consists of endocrinology, nutrition and surgery consultations, usually lasting 30 minutes every 6 months. These consultations usually include a physical exam (weight, height) and personalized diet/lifestyle recommendations. The Treatment as usual intervention is common to the Apolo_Bari Steppped-care intervention group and the treatment as usual control groups.
  Interventions: Other: Treatment as Usual for Bariatric Surgery

INTERVENTIONS:
Behavioral: Apolo_Bari Stepped-care intervention — Step 1 - Low-intensity intervention that will run on a private Facebook® group. Weekly, a subtopic and related activities are posted as short text/images. Patients are encouraged to participate by viewing publications, commenting, and posting their content.
  Step 2 - Will consist of an adjusted version of the Cognitive Behavior Treatment (CBT) program developed by Conceição et al. (2016). The intervention will last for 12-months and be delivered online by Facebook's functionalities, namely chat and calls. The intervention offered includes three components: 1) a psychoeducational cognitive-behavioral-based self-help manual that consists of 12 different modules. Each month a different topic will be covered and divided into four weekly sub-topics, which are supported with a set of related CBT tasks; 2) interactive call sessions with a psychologist (30 min at the beginning of each month); 3) monthly monitoring of risk-behaviors responded every session.
  Arms: Apolo_Bari Stepped-care intervention group
Other: Treatment as Usual for Bariatric Surgery — Treatment as Usual for bariatric surgery in portuguese public hospitals.
  Arms: Treatment as usual group

SUMMARY:
Bariatric surgery is the most effective treatment for severe obesity, yet a significant percentage of patients achieve suboptimal results or present long-term weight regain. Given the strong association between poor outcomes and post-surgery psychological factors, it is crucial to implement post-surgical psychological interventions.

This randomized controlled trial aims to compare the efficacy of a novel, cost-effective, and timely-personalized treatment delivering strategy (stepped-care) with two different intensities 1) low-intensity intervention delivered by Facebook®, and 2) high-intensity program delivered online. It is also intended to study predictors, outcome moderators/mediators, and the underlying mechanisms of weight regain. Participants' assessment will include measures of pathological eating behavior, psychological impairment, negative urgency, and emotional regulation.

DETAILED DESCRIPTION:
This research project intends to examine the effectiveness of a Cognitive Behavioral Therapy and psychoeducational based stepped-care program delivered online for patients submitted to bariatric surgery: APOLO_Bari. Therefore, a randomized controlled trial will compare a control group receiving multidisciplinary medical treatment as usual (TAU) for bariatric surgery in public health care centers in Portugal, and an intervention group receiving TAU plus the stepped-care APOLO-Bari web-based intervention.

The stepped-care APOLO-Bari intervention was designed to optimize weight loss, and prevent weight regain after bariatric intervention, promoting the adoption of healthy eating habits and lifestyle behaviors.

All participants will be assessed at baseline, 6- and 12- months after the beginning of the intervention, at the end of the 18-months intervention and at 6-months follow-up. Additionally, throughout the entire intervention, patients will respond to a short monthly monitoring questionnaire (MMQ) which consist of a self-monitoring online tool that allows patients to regularly input monitoring information regarding key disordered eating behaviors and their weight, maintaining a log of the individual process. Based on this information, a decision rule will be used to move patients through the different levels of interventions: Step 1: all patients receive intervention; Step 2: patients reporting at least one disordered eating behavior (e.g. grazing, binge-eating, skipping meals), or 2kg weight regain since the beginning of the intervention. If/when a patient moves to a new step of the protocol, the same set of measures will be responded before, in the middle, and at the end of that intervention.

ANOVAS for repeated measures and General Estimating Equations will be used to explore the differences between the groups in the various moments of evaluation. Hierarchical Linear Models with growth curves for repeated measurements will be used to explore the weight trajectories of patients in the two groups and to test predictors of weight variations. The PROCESS macro for SPSS will test moderators/mediators of the relationship between psychological variables, disordered eating behaviors, and weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Underwent Roux-en-Y Gastric Bypass or Gastric Sleeve
* Be at least 12 months after surgery;
* Have a Facebook® account and regular Internet access.

Exclusion Criteria:

* Under weight-loss medications;
* Having acute psychiatric or medical problems;
* pregnancy or lactation;
* illiteracy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Body max index | Change from Baseline (before the intervention), to 6-,12-, and 18-months (end of treatment) after baseline, and 6 months after end of treatment. Specific duration of time over which participant is assessed: 24 months.
  Calculated by WHO guidelines
Change in Disordered eating behaviors | Change from Baseline (before the intervention), to 6-,12-, and 18-months (end of treatment) after baseline, and 6 months after end of treatment. Specific duration of time over which participant is assessed: 24 months.
  Questionnaire developed for this study to evaluate the presence of key disordered eating behaviors (LOCE, binge-eating, grazing, and skipping meals). Higher scores indicate a higher presence of these problems.
Change in Grazing behavior | Change from Baseline (before the intervention), to 6-,12-, and 18-months (end of treatment) after baseline, and 6 months after end of treatment. Specific duration of time over which participant is assessed: 24 months.
  Repetitive Eating Questionnaire (Repeat-Q) - measure that assesses feelings, behaviors, and cognitions related to episodes of grazing resulting in two subscales: compulsive, and non-compulsive grazing. Higher scores indicate a higher presence of these problems.
Change in Eating disorder psychopathology | Change from Baseline (before the intervention), to 6-,12-, and 18-months (end of treatment) after baseline, and 6 months after end of treatment. Specific duration of time over which participant is assessed: 24 months.
  Eating Disorder_15 (ED-15) - measure that evaluates eating disorder psychopathology with subscales for weight and shape concerns and for eating concerns. Higher scores indicate a higher presence of these problems.
Change in Loss of control over eating | Change from Baseline (before the intervention), to 6-,12-, and 18-months (end of treatment) after baseline, and 6 months after end of treatment. Specific duration of time over which participant is assessed: 24 months.
  The Loss of Control over Eating Scale (LOCES) - measure that assesses the degree of LOC over eating in three aspects: behavioral, cognitive/dissociative and positive/euphoric. Higher scores indicate a higher presence of these problems.
Change in Difficulties in emotion regulation | Change from Baseline (before the intervention), to 6-,12-, and 18-months (end of treatment) after baseline, and 6 months after end of treatment. Specific duration of time over which participant is assessed: 24 months.
  Difficulties in Emotion Regulation Scale (DERS) - measure that assesses clinically relevant difficulties in emotion regulation through six dimensions: nonacceptance of emotional responses, difficulties engaging in goal-directed behavior when distressed, impulse control difficulties, lack of emotional awareness, limited access to effective emotion regulation strategies, and lack of emotional clarity. Higher scores indicate a higher presence of these problems.
Change in Negative urgency | Change from Baseline (before the intervention), to 6-,12-, and 18-months (end of treatment) after baseline, and 6 months after end of treatment. Specific duration of time over which participant is assessed: 24 months.
  UPPS-NU: Measure that assesses an individual's tendency to surrender to strong impulses, particularly under situations of negative emotions. Higher scores indicate a higher presence of these problems.
Change in Psychological impairment | Change from Baseline (before the intervention), to 6-,12-, and 18-months (end of treatment) after baseline, and 6 months after end of treatment. Specific duration of time over which participant is assessed: 24 months.
  Depression Anxiety Stress Scales (DASS) - measure that evaluates three dimensions: anxiety, depression, and stress. Higher scores indicate a higher presence of these problems.

SECONDARY OUTCOMES:
Satisfaction with intervention | Assessment at 18 months after the beginning of the intervention (End of treatment).
  Satisfaction questionnaire - measure developed to this study to addresses the utility and feasibility of the program from the patient's perspective. Higher scores indicate a higher satisfation with the program.
Attendance to the intervention. | Assessment at 18 months after the beginning of the intervention (End of treatment).
  Number of interactions on Facebook® private group, number of sessions attended, and number of monthly monitoring questionnaires responded.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar Universitário do Porto, Porto, Portugal